CLINICAL TRIAL: NCT00472797
Title: A Randomized, Multicenter, Two-arm, 12 Week Phase IIIb Study to Evaluate Quality of Life (QOL) Measures in Subjects With Relapsing Forms of Multiple Sclerosis (MS) Who Are Transitioning From Rebif® (Interferon Beta-1a) to Rebif New Formulation (RNF)
Brief Title: Rebif New Formulation (RNF) Quality of Life (QOL) Study
Acronym: RebiQoL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Ahmad Al-Sabbagh, Vice President Medical Affairs, US Neurology, EMD Serono, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27955
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Relapsing Multiple Sclerosis

ARMS (2):
- 1 (Active Comparator): Rebif New Formulation - Non Titrated
  Interventions: Drug: Rebif New Formulation Non Titrated
- 2 (Active Comparator): Rebif New Formulation - Titrated
  Interventions: Drug: Rebif New Formulation Titrated

INTERVENTIONS:
Drug: Rebif New Formulation Non Titrated — human interferon beta 1a - Rebif New Formulation
  Arms: 1
Drug: Rebif New Formulation Titrated — Human interferon beta 1a Rebif New Formulation
  Arms: 2

SUMMARY:
To evaluate the impact on Quality of Life (QOL), tolerability, treatment satisfaction, and injection site redness Rebif treated subjects with relapsing forms of MS who transition to a new formulation of Rebif (RNF).

ELIGIBILITY:
Inclusion Criteria:

1. Subject with a relapsing form of MS; diagnosis of MS is in accordance with the McDonald criteria
2. Subject currently taking Rebif 44mcg tiw, and has been on this treatment for at least 6 months (24 weeks) prior to study enrollment
3. Subject currently using Rebiject II and 29 gauge needle
4. Subject is between 18 and 60 years old inclusive
5. Subject is able to read and understand English
6. Subject is willing to follow study procedures
7. Subject has given written informed consent and signed HIPAA
8. Female subjects must not be either pregnant or breast-feeding and must lack childbearing potential, as defined by either: i) Being post-menopausal or surgically sterile, or ii) Using a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study. (Confirmation required within 30 days prior to start of the study)

Exclusion Criteria:

1. Use of any other injectable medications on a regular basis during the week prior to the screening period or during the screening or treatment periods. Receiving a single injection for treatment or prophylaxis of a condition unrelated to the subject's multiple sclerosis or the subject's Rebif® therapy (e.g., receiving a influenza or pneumococcus vaccination) is acceptable
2. Subject receiving MS therapy in addition (i.e., combination therapy) to Rebif® within 3 months prior to study enrollment or at any time during study protocol.
3. Subjects who have previously been on Rebif New Formulation (RNF).
4. Subject with progressive forms of Multiple Sclerosis (MS).
5. Subject with history of any chronic pain syndrome.
6. Subject has any other disease apart from MS that could better explain the subjects signs and symptoms.
7. Subject has complete transverse myelitis or bilateral optic neuritis.
8. Subjects that use any investigational drug or experimental procedure within 12 weeks of visit 1.
9. Subject received oral or systemic corticosteroids or ACTH within 30 days of visit 1 (prior to enrollment).
10. Subject has inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or alkaline phosphatase > 2.5 times the upper limit of the normal values.
11. Subject has inadequate bone marrow reserve, defined as a white blood cell count less than 0.5 x lower limit of normal.
12. Subject suffers from other current autoimmune disease.
13. Subject suffers from major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
14. Subject is pregnant or attempting to conceive
15. Visual or physical impairment that precludes completion of diaries and questionnaires.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dangond, MD, Study Director — EMD Serono
Locations (1):
- EMD Serono, Inc., Rockland, Massachusetts, United States

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 232 subjects were recruited from 25 Multiple Sclerosis (MS) Clinics in the US from April 2007 through November 2007.
Pre-assignment Details: Run-in period (up to 30 days) on Rebif® 44 mcg tiw: The run-in period included a Screening Visit; assessments consisted of informed consent, medical/disease history, physical exam and laboratory assessments which were performed in the two-week period prior to Study Day 1, (prior to the first dose of a new formulation of rebif)
Groups:
- New Formulation of Rebif - Non-Titrated: The new formulation of rebif is not approved and under investigation in the US
- New Formulation of Rebif - Titrated: The new frmulation of rebif is not approved and under investigation in the US
Period: Overall Study
Arm/Group | New Formulation of Rebif - Non-Titrated | New Formulation of Rebif - Titrated
Started | 119 | 113
Completed | 115 | 112
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Formulation of Rebif - Non-Titrated | New Formulation of Rebif - Titrated | Total
Number analyzed (Participants) | 119 | 113 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 119 | 113 | 232.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.0) | 42.8 (9.4) | 43.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 89 | 180.0
  Male | 28 | 24 | 52.0
Region of Enrollment [Number; unit: participants]
  United States | 119 | 113 | 232.0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Global Side Effects (GSE) on Multiple Sclerosis Treatment Concerns Quesionnaire (MSTCQ)
Description: The MSTCQ Global Side Effect domain assesses the degree of satisfaction on global side effect questions 9, 10 & 11 on a scale from 3 (not at all satisfied) to 15 (extremely satisfied). Percent change calculated as 100% * (score at week 12 - score at baseline) / score at baseline.
Time Frame: % change from Baseline to Week 12
Population: Safety: This population includes all subjects who received at least one dose of study drug. To explain difference in number, 1 subject lost to follow-up, 1 subject withdrew consent
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- All New Formulation of Rebif Subjects: All subjects combined in Intent to Treat (ITT) Population
Arm/Group | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 230
percent change | 5.0 (17.7)
Statistical Analysis 1: Comparison: All New Formulation of Rebif Subjects; A one-sided paired t-test across all subjects by combining the titrated and non-titrated new formulation groups was performed; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — P-Value denotes percent change from baseline to week 12 for all combined subjects; mean = 2.73, 97.5% CI [2.73 to 2.73]

2. Secondary Outcome: Total Score for Global Side Effects on Multiple Sclerosis Treatment Concerns Questionnaire (MSTCQ)
Description: The MSTCQ Global Side Effect domain assesses the subjects degree of satisfaction on global side effect questions 9, 10 & 11 on a scale from 3 (not at all satisfied) to 15 (extremely satisfied).
Time Frame: Baseline and Week 12
Population: Intent to Treat (ITT) and Last Observation Carried Forward (LOCF) Higher scores indicate a more favorable response
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Non-Titrated; Titrated: New formulation of rebif
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 117 | 113 | 230
score on scale
  Mean GSE at Baseline | 13.4 (1.7) | 13.4 (1.8) | 13.4 (1.7)
  Mean GSE at Week 12 (LOCF) | 14.0 (1.6) | 13.8 (1.6) | 13.9 (1.6)
  Percent Change - Baseline to Week 12 (LOCF) | 5.5 (16.5) | 4.5 (18.8) | 5.0 (17.7)
Statistical Analysis 1: Comparison: Non-Titrated vs Titrated; Test type: Superiority or Other; p = 0.466, ANOVA — P-value denotes difference between treatment groups
Statistical Analysis 2: Comparison: Non-Titrated; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — P-value denotes the mean percent change from baseline to week 12
Statistical Analysis 3: Comparison: Titrated; Test type: Superiority or Other; p = 0.003, t-test, 1 sided — P-value denotes the mean percent change from baseline to week 12

3. Secondary Outcome: Change in Score From Baseline to Week 12 for All Domains Other Than Global Side Effects on Multiple Sclerosis Treatment Concerns Questionnaire (MSTCQ)
Description: The MSTCQ in all domains assesses quality of life. The score for all domains other than the Global Side Effect ranges from 17 (most favorable) to 85 (least favorable). Change calculated as (score at week 12 - score at baseline.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 117 | 113 | 230
score on scale
  Injection System Satisfaction Domain | -3.2 (4.0) | -2.9 (4.1) | -3.1 (4.1)
  Side Effects Domain | -3.3 (6.4) | -2.3 (5.7) | -2.8 (6.1)
  Flu-Like Systems Domain | -0.9 (3.6) | -0.8 (3.6) | -0.8 (3.6)
  Injection Site Reactions Domain | -1.9 (3.2) | -1.3 (2.9) | -1.6 (3.1)
  Total Scores in all above Domains | -6.7 (8.8) | -5.3 (7.6) | -6.0 (8.3)
Statistical Analysis 1: Comparison: All New Formulation of Rebif Subjects; Change in total score from baseline to week 12 for all subjects combined. Lower scores indicate a more favorable response; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — P-value refers to change in total score from baseline to week 12 for all domains, except global side effect score, in the MSTCQ for all subjects combined; Paired t-test for change from baseline to week 12
Statistical Analysis 2: Comparison: Non-Titrated vs Titrated; Analysis evaluated differences between treatment groups in change in total score from baseline to week 12 for all domains, except global side effect score, in the MSTCQ. Lower scores indicate a more favorable response; Test type: Superiority or Other; p = 0.110, ANOVA — P-value refers to differences between treatment groups in change in total score from baseline to week 12 for all domains, except global side effect score, in the MSTCQ

4. Secondary Outcome: Total Score on Short-Form McGill Pain Questionnaire (SF-MPQ): Change in Baseline to Wk 12
Description: The SF-MPQ assesses Tolerability of Pain with 15 questions to evaluate the type and severity of pain experienced 60 minutes after an injection of study drug. Scores range from 0 (no pain) to 45 (severe pain).
Time Frame: Baseline to Week 12
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 117 | 113 | 229
score on scale | 0.7 (3.4) | 1.1 (3.9) | 0.9 (3.7)
Statistical Analysis 1: Comparison: Non-Titrated vs Titrated; Analysis evaluates total score from baseline to week 12 for differences between each treatment group; Test type: Superiority or Other; p = 0.302, ANOVA — P-value refers to differneces in total score from baseline to week 12 between treatment groups

5. Secondary Outcome: Tolerability in Pain Using Visual Analog Scale (VAS)
Description: The SF-MPQ included a visual analog scale, ranging from 0 to 100 mm, on which subjects rate pain from no pain (0 mm) to worst possible pain (100 mm). A rating of <5 mm was considered pain-free.
Time Frame: Baseline to Week 12
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 119 | 113 | 232
Participants
  Baseline - No. of Subjects Pain Free | 51 | 48 | 101
  Week 12 - No. of Subjects Pain Free | 53 | 48 | 101

6. Secondary Outcome: Tolerability - Redness at Injection Site
Description: Change in Baseline to Week 12 Last Observation Carried Forward(LOCF)- A blinded assessment of injection site redness was conducted by a health care professional (1-72 hours) after the most recent injection measuring redness at its widest diameter in mm. Diameter of Redness, lower is better.
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 114 | 110 | 224
mm | -2.3 (27.7) | -3.1 (28.2) | -2.7 (27.9)
Statistical Analysis 1: Comparison: Non-Titrated vs Titrated; Analysis evaluates differences between treatment groups in change in diameter of injection site redness from baseline to week 12; Test type: Superiority or Other; p = 0.899, ANOVA — P-value denotes differences between treatment groups in change in diameter of injection site redness from baseline to week 12

7. Other Pre Specified Outcome: SF-36 Physical and Mental Component Scores
Description: Change from Baseline to each visit for Physical and Mental Component scores for SF-36. Score is norm-based with a mean of 50 and a standard deviation of 10.
Time Frame: Change from Baseline to Each Visit
Population: ITT
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Number analyzed (Participants) | 119 | 113 | 232
Score
  Physical Component Score - Baseline | 43.4 (9.4) | 43.6 (9.3) | 43.5 (9.3)
  Physical Component -Change from Baseline to Wk 12 | 1.8 (5.7) | 2.0 (4.3) | 1.9 (5.0)
  Physical Component -Change from Baseline to Wk 36 | -0.2 (7.7) | 1.5 (6.0) | 0.6 (7.0)
  Physical Component -Baseline to Ext. Visit 1 | 2.0 (6.5) | 1.7 (6.6) | 1.9 (6.5)
  Physical Component -Baseline to Ext Visit 3 | 1.0 (6.5) | 2.0 (6.4) | 1.5 (6.4)
  Physical Component -Baseline to Exit Visit/LOCF | 0.4 (6.4) | 1.4 (6.4) | 0.9 (6.4)
  Mental Component - Baseline | 46.1 (10.9) | 46.1 (10.9) | 46.1 (10.9)
  Mental Component - Change from Baseline to Week 12 | 2.5 (8.7) | 1.3 (9.1) | 1.9 (8.9)
  Mental Component - Change from Baseline to Week 36 | 1.8 (10.6) | -0.8 (10.0) | 0.5 (10.4)
  Mental Component - Baseline to Ext Visit 1 | 0.3 (10.7) | -1.2 (8.9) | -0.4 (9.8)
  Mental Component - Baseline to Ext Visit 3 | 1.3 (11.2) | 0.1 (10.4) | 0.7 (10.8)
  Mental Component - Baseline to Exit/LOCF | -0.1 (11.2) | 0.1 (9.7) | 0.0 (10.5)
Statistical Analysis 1: Comparison: All New Formulation of Rebif Subjects; Physical Component - Change from Baseline to Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired
Statistical Analysis 2: Comparison: All New Formulation of Rebif Subjects; Physical Component - Change from Baseline to Week 36; Test type: Superiority or Other; p = 0.234, t-test, 2 sided; Paired
Statistical Analysis 3: Comparison: All New Formulation of Rebif Subjects; Physical Component - Change from Baseline to Extension Visit 1; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Paired
Statistical Analysis 4: Comparison: All New Formulation of Rebif Subjects; Physical Component - Change from Baseline to Extension Visit 3; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; Paired
Statistical Analysis 5: Comparison: All New Formulation of Rebif Subjects; Physical Component - Change from Baseline to Exisit Visit LOCF; Test type: Superiority or Other; p = 0.036, t-test, 2 sided; Paired
Statistical Analysis 6: Comparison: All New Formulation of Rebif Subjects; Mental Component - Baseline to Week 12; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Paired
Statistical Analysis 7: Comparison: All New Formulation of Rebif Subjects; Mental Component - Baseline to Week 36; Test type: Superiority or Other; p = 0.468, t-test, 2 sided; Paired
Statistical Analysis 8: Comparison: All New Formulation of Rebif Subjects; Mental Component - Change from Baseline to Extension Visit 1; Test type: Superiority or Other; p = 0.602, t-test, 2 sided; Paired
Statistical Analysis 9: Comparison: All New Formulation of Rebif Subjects; Change from Baseline to Extension Visit 3; Test type: Superiority or Other; p = 0.414, t-test, 2 sided; Paired
Statistical Analysis 10: Comparison: All New Formulation of Rebif Subjects; Change from Baseline to Exit Visit LOCF; Test type: Superiority or Other; p = 0.991, t-test, 2 sided; Paired

ADVERSE EVENTS:
Arm/Group | Non-Titrated | Titrated | All New Formulation of Rebif Subjects
Serious Adverse Events (participants affected / at risk) | 10/118 | 6/113 | 16/231
Other Adverse Events (participants affected / at risk) | 90/118 | 78/113 | 168/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Non-Titrated (N=118) | Titrated (N=113) | All New Formulation of Rebif Subjects (N=231)
Artrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1/1 (1)
Cardiomiopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1/1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1/1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1/1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1/1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1/1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1/1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1/1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1/1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1/1 (1)
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1/1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1/1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1/1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1/1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1/1 (1)
Renal Artery Fibromuscular Dysplasia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1/1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1/1 (1)
Secondary Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1/1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1/1 (1)
Suicidal ideation (Social circumstances) | 1 (1) | 0 (0) | 1/1 (1)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0) | 1/1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Titrated (N=118) | Titrated (N=113) | All New Formulation of Rebif Subjects (N=231)
Chills (General disorders) | 9 (9) | 4 (4) | 13 (13)
Headache (Nervous system disorders) | 38 (38) | 28 (28) | 66 (66)
Influenza-like Illness (General disorders) | 11 (11) | 9 (9) | 20 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 1 (1) | 14 (14)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9) | 18 (18)
Pain (General disorders) | 20 (20) | 16 (16) | 36 (36)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 12 (12)
Urinary tract infection (Renal and urinary disorders) | 6 (6) | 9 (9) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor any Principal Investigators shall publish or present any results from such Study to any third parties until: (i) EMD Serono publishes the results from all sites participating in such Study; (ii) Institution receives notification from EMD Serono that publication of the multi-site results is no longer planned; or (iii) twenty-four (24) months following the completion of the multi-site study at all sites, whichever occurs first.